CLINICAL TRIAL: NCT02056574
Title: Phase 2, Multicenter Randomized, Double-Blind, Placebo-Controlled, Safety and Efficacy Study Evaluating a Single Dose of Intravenous NA-1 in Patients With Subarachnoid Hemorrhage Undergoing Endovascular Repair of Ruptured Intracranial Aneurysms
Brief Title: Safety and Efficacy Study of a Single Dose of NA-1 in Patients Undergoing Endovascular Repair of Ruptured Aneurysms
Acronym: ENACT-2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: NoNO Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA-1-006
Record Dates: First submitted 2014-02-04; First posted 2014-02-06 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-03

CONDITIONS: Subarachnoid Hemorrhage; Ruptured Intracranial Aneurysm
Keywords: Endovascular repair; Subarachnoid hemorrhage; Ruptured intracranial aneurysm; Stroke; Coiling; NA-1
MeSH Terms: conditions — Subarachnoid Hemorrhage; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NA-1 (Experimental): 20 amino acid peptide that consists of a 9 amino acid domain that inhibits PSD-95 and an 11 amino acid domain that enables the peptide to cross the blood-brain barrier. Single intravenous dose of 2.6 mg/kg of NA-1 administered as a 10-minute infusion.
  Interventions: Drug: NA-1
- Placebo (Placebo Comparator): Single intravenous dose of 2.6 mg/kg of placebo administered as a 10-minute infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NA-1
  Arms: NA-1
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single-dose study investigating the safety and efficacy of NA-1 in patients with subarachnoid hemorrhage (SAH) undergoing endovascular repair of ruptured intracranial aneurysms. Up to 300 male and female patients with SAH undergoing endovascular repair of a ruptured intracranial aneurysm will be dosed with 2.60 mg/kg of NA-1 or placebo as a 10 minute intravenous infusion after completion of the endovascular procedure on Day 1 of the study period. Subjects will undergo interim procedures at Day 2-4, Day 30-45, and end-of-study procedures on Day 90.

ELIGIBILITY:
Inclusion Criteria:

* 1. A diagnosis of a ruptured brain aneurysm deemed suitable for repair by neuroendovascular techniques involving intraluminal occlusion by detachable platinum coils, or any neuroendovascular technique such as balloon-assisted coiling, stenting, or flowed diversion.
* 2. Patient should be Grade II-IV on the WFNS grading scale for SAH.
* 3. Male or female with a minimum age of 18 years on the day of enrolment.
* 4. Female subjects of childbearing potential: Negative pregnancy test.
* 5. Non-surgically sterile males or males with partners of childbearing potential must be willing to use condoms with spermicide for 3 months after completion of dosing.
* 6. Body weight less than or equal to 180 kg.
* 7. Vital signs on admission:

  * Blood pressure between 80-180 mm Hg systolic/50-100 mm Hg diastolic;
  * Body temperature ≤ 38.5C.
* 8. Informed consent and availability of the subject for the entire study period and willingness of the subject to adhere to protocol requirements.

Exclusion Criteria:

* 1. Prior SAH within 6 months of presentation.
* 2. Dissecting or mycotic brain aneurysm.
* 3. Planned endovascular vessel sacrifice as the primary modality for aneurysm treatment.
* 4. Known history of life-threatening allergic reaction to any medication.
* 5. Chronic renal disease defined as a baseline serum creatinine > 150 µmol/L.
* 6. Women who are pregnant, or have a positive urine or blood (β-hCG) pregnancy test.
* 7. Women who are breastfeeding.
* 8. Any clinically significant psychiatric or psychological disease, which would preclude the patient from completing the protocol.
* 9. Pre-morbid (estimated) modified Rankin scale score of >1.
* 10. Previous major stroke.
* 11. Patients with known HIV infection.
* 12. Participation in a clinical trial with an investigational drug within 30 days preceding this study.
* 13. Previous participation in the ENACT trial (e.g, to treat a prior aneurysm), participation in another trial involving NA-1 or prior receipt of NA-1.
* 14. Any other medical condition that the site investigator deems would put the patient at excessive risk of participation in the study or an expected life expectancy less than 1 year or that would result in inability to collect clinical outcomes at 90 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2019-11 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) | 90 days
  Proportion of subjects achieving independent functioning as defined as a score of 0-1 on the mRS at Day 90.

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) | 30-45 days
  Proportion of subjects achieving a good outcome as defined as a score of 0-1 on the mRS at Day 30-45.
National Institutes of Health Stroke Scale (NIHSS) | 90 days
  Proportion of subjects achieving a good outcome as defined as a score of 0-1 on the NIHSS at Day 90.
Mortality | 90 days
  Rate of subarachnoid hemorrhage related mortality over the 90 day study period.
In-hospital length of stay | 90 days
  Duration of in-hospital length of stay.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tymianski, MD, PhD, Study Director — NoNO Inc.; Cameron G McDougall, MD, Principal Investigator — Barrow Neurological Institute; Michael D Hill, MD, Principal Investigator — Foothills Medical Centre
Locations (12):
- United States (5):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Colorado Neurological Institute, Englewood, Colorado
  - University of Michigan - Neurosurgery, Ann Arbor, Michigan
  - Oregon Health and Science University, Portland, Oregon
  - University of Wisconsin, Madison, Wisconsin
- Canada (7):
  - Foothills Medical Centre, Calgary, Alberta
  - QEII Health Sciences Centre - Halifax Infirmary, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Hopital de l'Enfant Jesus, Québec, Quebec